CLINICAL TRIAL: NCT01038050
Title: Study Effects of Ginkgo Biloba Extract on Endothelial Cell Function and Genetic Effects on the Response to Ginkgo Biloba Extract in Diabetic Patients With Stable Coronary Artery Disease
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Liang-Yu, Lin/ Attending phsician, Taipei Veterans General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VGHIRB 98-10-02
Record Dates: First submitted 2009-12-20; First posted 2009-12-23 (Estimated); Last update posted 2009-12-23 (Estimated); Status verified 2009-12

CONDITIONS: Type 2 Diabetes Mellitus; Coronary Artery Disease
Keywords: Endothelial progenitor cell; endothelial function(FMD); Gingko Biloba Extract; Type 2 Diabetes mellitus; Stable coronary artery disease; Endothelial progenitor cells Numbers
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Coronary Artery Disease | interventions — Ginkgo biloba extract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Ginkgo Biloba Extract (GBE) — Ginkgo Biloba Extract 40 mg 1# tid per day for 3 months(90 days)
  Other Names: Cerenin(Ginkgo Biloba Extract) film-coated 40 mg

SUMMARY:
Type 2 diabetes is associated with a markedly increased risk for atherosclerotic coronary arteries and cerebrovascular diseases. The major cause of death in diabetic patients is cardiovascular disease in the world including Taiwan. Atherosclerosis is a progressive disease characterized by the response of the vessel wall to chronic, multifactorial injury, which leads ultimately to the formation of atheromatous or fibrous plaques. Endothelial dysfunction is thought to be the initial stage of atherosclerosis. Endothelial dysfunction leads to impaired control of vascular tone, a decreased in the release of anti-inflammatory factors and reduced availability of nitric oxide. Endothelial dysfunction portends diabetic vasculopathy. The loss of intact endothelial integrity and function sets in motion a cascade of serial events that lead to atherosclerosis and cardiovascular complications.

The standard extracts of G. biloba leaves [G. biloba extract (GBE)] are now demonstrated the cardiovascular, cerebrovascular and neuroprotective effects. The mixture of biologically active ingredients in GBE accounts for the pleiotropic effects, including antioxidant effects, inhibition of platelet aggregation and thromboxane B2 production, vasodilation and modulation of cholesterol metabolism. Clinically, GBE was widely used in management of vertigo、dementia and improving peripheral circulation. In our previous study, ginkgo biloba extract inhibits tumor necrosis factor-alpha-induced reactive oxygen species generation, transcription factor activation, and cell adhesion molecule expression in human aortic endothelial cells. In addition, the similar benefit of prevention atherosclerosis was also found in animal study.

Heme oxygenase-1 (HO-1) is a factor associated with higher risk of developing some vascular disease and also a rate-limiting enzyme in heme degradation, leading to the generation of free iron, biliverdin, and carbon monoxide (CO). CO exerts potent antiproliferative and anti-inflammatory effects in the vascular walls, thereby influencing neointimal formation after vascular injury. In addition, biliverdin is subsequently metabolized to bilirubin by the enzyme biliverdin reductase. Therefore, induction of HO-1 elicits potent anti-inflammatory, antiproliferative, antithrombotic, and antioxidant effects in the circulation via the generation of CO and bilirubin. Interestingly, recent study found that a long guanidine thymidine dinucleotide repeat [(GT) n≧ 30] in the HO-1 promotor, which is linked to impaired inducibility, is associated with a higher frequency of vascular access failure.

In the present study, we will investigate the effect of GBE on recovering endothelial dysfunction and inflammation in diabetic patients with stable coronary artery disease. In particularly, we intend to determine whether the GBE modulates the HO-1 expression and investigate whose genotyping including some candidate gene about atherosclerosis and hypertension will have most therapeutic effect of GBE.

ELIGIBILITY:
Inclusion Criteria:

* Thirty type 2 diabetes mellitus with stable coronary disease
* Aged 18-80 year-old

Exclusion Criteria:

* Previous underwent coronary artery bypass surgery or percutaneous angioplasty
* Under insulin injection patients
* Renal or hepatic function impairment
* Pregnant women
* Poor BP control(BP>175/105 mmHg)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2009-10; Primary Completion 2010-11 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Number of endothelial progenitor cells, endothelial function(FMD) | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Jaw-Wen Chen, MD, Principal Investigator — Division of Cardiology, Taipei Veterans General Hospital; Chin-Chou Huang, MD, Principal Investigator — Division of Cardiology, Taipei Veterans General Hospital
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan